CLINICAL TRIAL: NCT00090207
Title: A Randomized, Double-Blind, Parallel-Group Study Conducted Under In-House Blinding Conditions to Determine the Safety, Tolerability and Efficacy of Aprepitant Regimen Compared to Ondansetron Regimen for the Prevention of Chemotherapy Induced Nausea and Vomiting (CINV) Associated With High Dose Cisplatin in Cycle 1
Brief Title: Aprepitant for the Prevention of Chemotherapy Induced Nausea and Vomiting (CINV) Associated With Highly Emetogenic Chemotherapy (0869-801)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0869-801; 2004_005
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0869, aprepitant / Duration of Treatment: 3 days
Drug: Comparator: ondansetron / Duration of Treatment: 4 days

SUMMARY:
A multicenter trial to assess the safety and efficacy of an investigational drug in the prevention of chemotherapy-induced nausea and vomiting (CINV) in patients with confirmed solid tumors who will be treated with a chemotherapy regimen that includes cisplatin. The study will evaluate the investigational drug for the treatment of CINV during the first cycle of treatment with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than 18 years of age.
* Patient is scheduled to receive his/her first

course of cisplatin chemotherapy for a solid tumor.

* Patient has a prognosis (life expectancy) greater than or equal to 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2004-01-13 (Actual); Primary Completion 2004-09-30 (Actual); Study Completion 2004-09-30 (Actual)

PRIMARY OUTCOMES:
Patient vomiting

SECONDARY OUTCOMES:
Number of rescue therapies

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Schmoll HJ, Aapro MS, Poli-Bigelli S, Kim HK, Park K, Jordan K, von Pawel J, Giezek H, Ahmed T, Chan CY. Comparison of an aprepitant regimen with a multiple-day ondansetron regimen, both with dexamethasone, for antiemetic efficacy in high-dose cisplatin treatment. Ann Oncol. 2006 Jun;17(6):1000-6. doi: 10.1093/annonc/mdl019. Epub 2006 Mar 8. PMID 16524979
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/policies-perspectives.html